CLINICAL TRIAL: NCT06181188
Title: The Use of Ketamine for Conscious Sedation in Flexible Bronchoscopy
Brief Title: Use of Ketamine for Conscious Sedation in Flexible Bronchoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jess T. Anderson, Pulmonary & Critical Care Fellow, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: C.2019.050
Record Dates: First submitted 2019-12-10; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Conscious Sedation; Patient Satisfaction; Ketamine
Keywords: Conscious Sedation; Bronchoscopy; Ketamine
MeSH Terms: conditions — Patient Satisfaction | interventions — Ketamine; Midazolam; Fentanyl

STUDY DESIGN:
Intervention Model Description: Single blinded randomized control trial. The control arm will receive a combination of midazolam and fentanyl. The study arm will receive a combination of midazolam and ketamine.
Who Masked: Participant
Masking Description: Envelops with pre-randomized and documents will be sealed and placed in a locked cabinet. Once a patient has been enrolled an envelop will be obtained indicating which arm the patient will be enrolled into. The study drugs will be labeled A (ketamine), B (midazolam), and C (fentanyl) and will be referred to as A, B, or C during the procedure to as to maintain anonymity from the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketamine and Midazolam (Experimental): Patients will receive 1mg of midazolam and a bolus of 0.25 - 0.5mg/kg of ketamine to initiate sedation. Additional 10-20mg of ketamine will be given every 3-5 minutes to achieve adequate sedation. If additional anxiolysis is needed, additional doses of midazolam will be given every 3-5 minutes in 1mg increments. .
  Interventions: Drug: Ketamine; Drug: Midazolam
- Midazolam and Fentanyl (Active Comparator): Patient will receive midazolam and fentanyl in 1mg and 25mcg increments respectively until adequate procedural sedation is achieved. Additional increments will be given every 3-5 minutes as needed to achieve adequate sedation.
  Interventions: Drug: Midazolam; Drug: Fentanyl

INTERVENTIONS:
Drug: Ketamine — Patients will receive a combination of ketamine and midazolam for conscious sedation
  Other Names: Ketalar
  Arms: Ketamine and Midazolam
Drug: Midazolam — Patients will receive 1mg of midazolam regardless of which arm they are in and my be given 1mg doses for added sedation as needed every 3-5 minutes
  Other Names: Versed
Drug: Fentanyl — Patients randomized to the midazolam and fentanyl arm will receive 25mcg incremental doses for procedural sedation
  Arms: Midazolam and Fentanyl

SUMMARY:
In this study, the investigators plan to conduct a single blinded randomized controlled trial in the Pulmonary Service to demonstrate the efficacy of ketamine and its utility in moderate sedation. Patients presenting for bronchoscopy who meet inclusion criteria will be approached, and if amenable, will be consented and enrolled. Patients will be randomized to receive either 1 mg of midazolam and ketamine 0.25 to 0.5 mg/kg loading dose with subsequent doses of 10-20 mg IV or standard fentanyl and midazolam in 25mcg and 1mg increments respectively for moderate sedation during their procedure. The primary outcome will be patient satisfaction, which will be measured a using patient clinical satisfaction form. A number of secondary outcomes will include the following: (1) provider satisfaction (2) the time from sedation administration to procedure start (when the scope is inserted), (3) the time from sedation to scope removal from the trachea (4) the time from sedation to discharge (defined as the time from the end of the procedure until the patient meets discharge criteria from the recovery area), (5) total dose of medications given (including midazolam, fentanyl, and ketamine), (6) adverse events, (7) vital signs, (8) and the need for additional medications, in particular reversal agents.

DETAILED DESCRIPTION:
The investigators propose to carry out a single blinded randomized controlled trial where 33 patients will receive midazolam and ketamine for sedation in one arm and 33 will receive the standard fentanyl and midazolam combination in the other arm. During the procedure, the investigators will measure and record vital signs as well as the total dose of medication used. After the procedure, the investigator will note the time to recovery and discharge. The bronchoscopist will be asked to assess the quality of the procedure as well as a checklist to the patient to be done immediately after the procedure and 48 hours post procedure.

A patient presents to the pulmonary clinic for a scheduled outpatient bronchoscopy. During the initial visit to discuss the need for bronchoscopy, patients will be provided with a brochure on the study and advised that if they meet inclusion criteria, they may elect to participate. If the patient elects to participate in the study and meets inclusion and exclusion criteria they will be consented and enrolled. Once enrolled, the study personnel will then retrieve the subject's assigned envelope that will contain all the data collection forms and the study medication will be ordered. If the patient is enrolled in the ketamine arm, an order for ketamine will be placed in in the electronic medical record to the inpatient OR pharmacy for 10mg/ml (10ml) prefilled syringe. Pulmonary clinic nursing personnel will pick up the ketamine syringe from inpatient OR pharmacy. In the Bronchoscopy Suite, nurse will affix a sticker "Drug A" to cover the ketamine 10mg/mL pharmacy label. The remainder of the medications will be pulled from the pyxis machine in the bronchoscopy suite and kept on standby by the bedside nurse.

Once consented, the nurse or physician taking care of the patient will then take the sealed envelope within the packet containing the subject's randomized medication assignment and give this sealed envelope to the nurse involved in the subject's care to retrieve the medication. To maintain the study protocol the ketamine syringe will be labeled as 'drug A" The bedside nurse will label the syringe with midazolam and fentanyl as "drug B and drug C" respectively along with the amount, the patient name and the initial of the preparer, then give the medications to the attending physician for verification and administration by either the attending physician or fellow physician under direct supervision of the attending physician. The patient will be blinded to the study medication but the physicians and nursing staff will know the identity of the medications being administered. The subject will continue on with care as directed by the provider. There will be at least two licensed providers in the room for the duration of the procedure.

In regards to quality of sedation, procedural sedation will be titrated to achieve a RASS score of negative 1 to negative 3. In the patient's randomized to the ketamine arm they will receive an initial 1mg dose of IV midazolam for anxiolysis followed by Ketamine at an initial dose of 0.25 - 0.5 mg/kg administered over 1 minute. Additional doses of ketamine 10-20mg will be administered every 5-10 minutes until an appropriate level of sedation is achieved. Additional midazolam can be given for anxiety at the discretion of the attending physician. If the procedure calls for fentanyl to be used instead of ketamine, midazolam will be given in 1mg and fentanyl in 25mcg increments every 3 minutes and titrated to achieve a RASS of -3. During the procedure, the physician and nursing staff will refer to ketamine as "A" and then the dose (e.g. "please administer 10 mg of A") and midazolam as "B" in order to prevent the subject from knowing the identity of the study medication. If the bronchoscopist does not feel adequate sedation has been achieved after several doses of ketamine (at least 4 doses), they may convert the procedure to standard sedation consisting of fentanyl and midazolam and drop the subject from the study. Additionally, if the procedure is started and it is determined that the patient cannot be adequately sedated then the physician can elect to abort the procedure and drop the subject from the study. After completion of the procedure, the bronchoscopist will be given a form in which to rate the quality of procedural sedation; attached for review. During the procedure, vital signs and medication dose administration data will be recorded on the medication use sheet as already used in the BAMC pulmonary suite. Following the procedure, all immediate complications during the procedure will be recorded.

The investigator will record the time elapsed from medication administration until discharge from the recovery area. Subjects will be discharged from the recovery area after they meet preset parameters found in the standard operating procedures of the bronchoscopy suite. Procedural times such start time, completion of procedure, and total dose of sedation will be documented in the procedural report as currently preformed for all bronchoscopies. The total dose of sedation will be added to the procedural report by a study team member after the physician has filled out the report and submitted their sedation checklists as detailed below in order to maintain proper blinding. Immediately following the procedure, the bronchoscopist will complete a form rating: the overall quality of sedation, rating of subject discomfort, sedation-related technical difficulties, and depth of sedation. It will also me noted on the data recording form if the patient has an active prescription for opioids, benzodiazepines, or if they consume greater than or equal to five alcohol drinks per week.

After the subject meets the preset parameters found in the standard operating procedures of the bronchoscopy suite for discharge, a post-procedural checklists will be administered and the subject will be discharged home. The subject will be contacted via phone 48 hours after the procedure and will be asked to rate the quality of the procedure via the modified PSSI index as well as additional questions about their oral intake and if they experienced any side effects specific to ketamine. A sample of the script for the post-procedural phone call will be attached for review. The investigator will attempt to contact each subject at least 3x starting 48 hours after the procedure for two more days. voicemails will be left after each attempt. If they are unreachable, they will then be noted as lost to follow up.

All checklists will be sealed into separate envelopes and will be placed in the subject's overall study envelope. The envelopes will remain sealed until the study results are analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 to 75 years who present to the pulmonary clinic for bronchoscopy and considered for airway survey, transbronchial biopsy, endobronchial biopsy, or bronchoalveolar lavage.
* Provider performing the bronchoscopy

Exclusion Criteria:

* Systolic blood pressure over 180mmHg and/or diastolic blood pressure over 110 on two consecutive readings
* Tachycardia greater than 120 beats/minute on two consecutive measurements
* Any allergy to ketamine, fentanyl, or midazolam
* Patient is pregnant or refuses pregnancy test,in women of child-bearing potential*
* American Society of Anesthesiologists (ASA) score > 3
* Presence of a history of psychosis, hallucinations, and/or a psychotic disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Patient sedation satisfaction with sedation instrument | A survey will be conducted upon the completion of the procedure.
  A twenty one question survey assessing patient satisfaction using a 7-point Likert Scale. A "1" on the scale would indicated very satisfied, 2 - satisfied, 3 - somewhat satisfied, 4 - neither satisfied nor dissatisfied, 5 - somewhat dissatisfied, 6 - dissatisfied, and 7- very dissatisfied.
Patient sedation satisfaction with sedation instrument | A follow up survey will be conducted 24-48 hours after the completion of the bronchoscopy. The average of both survey's will then be used to score the overall satisfaction of sedation.
  A twenty one question survey assessing patient satisfaction using a 7-point Likert Scale. A "1" on the scale would indicated very satisfied, 2 - satisfied, 3 - somewhat satisfied, 4 - neither satisfied nor dissatisfied, 5 - somewhat dissatisfied, 6 - dissatisfied, and 7- very dissatisfied.

SECONDARY OUTCOMES:
Clinician satisfaction with sedation instrument | Upon completion of the procedure
  A twenty one question survey assessing patient satisfaction using a 7-point Likert Scale. A 1 indicates very satisfied, 2 - satisfied, 3 - somewhat satisfied, 4 - neither satisfied nor dissatisfied, 5 - somewhat dissatisfied, 6 - dissatisfied, and 7- very dissatisfied.
time from sedation administration to procedure start | during the procedure
  time for when the initial sedation is given to when the scope is inserted
procedural time | during the procedure
  Time from when sedation is given to when the scope is removed from the airway
Total time | during the procedure
  Time from when sedation is first given to when the patient meets discharge criteria
Total dose of medications given | during the procedure
  Total amount of medication given, ketamine will be measured in milligrams (mg), versed in mg, and fentanyl in micrograms with total dose of each calculated, direct comparison will not be possible however will allow clinicians to evaluate relative sedatives used.
Blood pressure | during the procedure
  Blood pressure - measured in mmHg
Heart Rate | during the procedure
  measured in beats per min (BPM)
Oxygen Saturation | during the procedure
  measured as SPo2
End Tidal Co2 | during the procedure
  measured in mmHg
Respiratory Rate | during the procedure
  measured as the number of breaths per minute

OTHER OUTCOMES:
A patient's history of alcohol consumption. | at enrollment and during the procedure
  The amount of alcoholic drinks consumed on a daily basis. The amount of sedating medication will then be recorded and a comparison will be made between patients who actively use alcohol to those who do not.
A patient's history of chronic opioid use. | at enrollment and during the procedure
  The amount of opioids used if patient has a current prescription for opioids. The amount of sedating medication will then be recorded and a comparison will be made between patients who actively use opioids to those who do not.
A patient's history of chronic benzodiazepine use. | at enrollment and during the procedure
  The amount of benzodiazepines will be recorded. The amount of sedating medication will then be recorded and a comparison will be made between patients who actively use benzodiazepines to those who do not.

CONTACTS AND LOCATIONS:
Overall Officials: Jess Anderson, DO, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No